CLINICAL TRIAL: NCT05411224
Title: Investigation of the Effect of Custom Made Insoles on Foot Sole Pressure Distribution and Gait Parameters in Patients With Morton's Neuroma
Brief Title: Investigation of the Effect of Custom Made Insoles on Foot Pressure Distribution and Gait Parameters in Patients With Morton's Neuroma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Özlem Feyzioğlu, Asistant Professor, Acibadem University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-2909
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Morton Neuroma
MeSH Terms: conditions — Morton Neuroma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Morton Nuroma (Experimental): In patients with Morton Neuroma, stride length, stance phase percentage, swing phase percentage, cadence and speed parameters, and fore, mid and hind foot pressure distribution will be recorded with the Zebris FDM-THM-S treadmill system in the analysis of barefoot walking after the physical examination evaluation of the cases.
  Interventions: Other: Custom made orthosis

INTERVENTIONS:
Other: Custom made orthosis — In patients with Morton Neuroma, stride length, stance phase percentage, swing phase percentage, cadence and speed parameters, and fore, mid and hind foot pressure distribution will be recorded with the Zebris FDM-THM-S treadmill system in the analysis of barefoot walking after the physical examination evaluation of the cases.While the treadmil is in a static state, pressure distribution measurement will be taken by baropedography, and personalized insoles will be produced according to the baropedographic pressure map. Patients will be delivered to the patient for indoor and outdoor use for 4 weeks. After a 4-week usage period, measurements related to pressure and walking parameters will be repeated.

SUMMARY:
The aim of our study is to investigate the effect of the use of custom made insoles in the treatment of Morton's neuroma on foot pressure, temporal and spatial gait parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral Morton neuroma
* Confirmation of the diagnosis of Morton's neuroma with Magnetic Resonance Imaging (MRI)
* Pain level of the patients while walking is at least 3 according to the Visual Analogue Scale (VAS).
* Volunteer to work

Exclusion Criteria:

* Symptomatic musculoskeletal disease in the lower extremity
* Peripheral nervous system disease
* Presence of rigid deformity in the foot
* Extremity or contralateral extremity surgery with Morton's neuroma

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Step length (centimeter- cm) | 4weeks
  Step length (cm) will be evaluated by Zebris (Zebris Medical Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Aim of the system analyzes gait of the patients. Step length describes the distance between the heel contact of one side of the body and the heel contact of the contralateral side.
Stance phase percentage (%) | 4 weeks
  Stance phase percentage (%) will be evaluated by Zebris (Zebris Medical Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Stance phase percentage describes the phase of a gait cycle in which the foot has contact with the ground.The unit is expressed as a percentage.
Swing phase percentage (%) | 4 weeks
  Swing phase percentage (%) will be evaluated by Zebris (Zebris Medical Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Swing phase describes the phase of a gait cycle during which the foot has no contact with the ground. The unit is expressed as a percentage
Cadance | 4 weeks
  Cadence (steps/min) will be evaluated by Zebris (Zebris Medical -Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. Cadence is steps/minute. It is defined as the step frequency.
Velocity | 4 weeks
  Velocity will be evaluated by Zebris (Zebris Medical -Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. The system measures average gait speed during the analyzed measuring interval. The unit is expressed as km/hr.
Foot pressure distiribution | 4 weeks
  Foot pressure distiribution will be evaluated by Zebris (Zebris Medical -Limited -, Germany) FDM (Force distribution measurement ) System. Participants will walk barefoot on the Zebris FDM (Zebris Medical Limited, Germany) treadmill system. The system evaluate the average maximum values reached in N/cm² for the three zones: toes, mid-foot and heel.
Pain - Visual Analogue Scale | 4 weeks
  Visual Analogue Scale is one of the simple and common methods used in pain assessment. Self reported pain intensity during the rest and the activity measured by 0-10 centimeter chart. Visual Analogue Scale (VAS), where 0 indicates no pain or best and 10 indicates the most intense pain imaginable or worst. The patient will mark the severity of the pain on a 10 cm long chart.

CONTACTS AND LOCATIONS:
Overall Officials: Selim Muğrabi, MD, Principal Investigator — Fulya Foot Surgery Clinic
Locations (1):
- Fulya Foot Surgery, Istanbul, Turkey (Türkiye)